CLINICAL TRIAL: NCT06531720
Title: Comparison of the Effects of Mucosa Tissue Healing in Patients Wearing a Removable Prosthetic Restoration - Pilot Study.
Brief Title: Comparison of the Effects of Oral Ulceration Healing in Patients Wearing a Removable Denture
Acronym: MUCOSA HEALING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUM MUCOSA HEALING
Record Dates: First submitted 2024-07-12; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Oral Mucosa; Ulcer
Keywords: prosthetic materials; functional properties; antibacterial properties; chlorhexidine; choline salicylate
MeSH Terms: conditions — Oral Ulcer | interventions — chlorhexidine gluconate; choline salicylate; Gels; Control Groups

STUDY DESIGN:
Intervention Model Description: According to randomization patients suffering from oral mucosa lesion (OML) were divided into three groups:
  * Group I: oral mucosa lesions treated with 0,2% CHX topical use,
  * Group II: oral mucosa lesions treated with 8,7% CHS topical use and
  * Group III: oral mucosa lesions as control group-CON with no specific OML treatment.
  The efficacy of oral topical medications in aiding regeneration and healing of oral soft mucosa, caused by the use of removable prosthetic restorations was analyzed. The evaluation of the efficacy of these agents was based on a comparison of the area of OML before and after the treatment. Patients in the control group were not using any topical medication.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A randomized, double-blind study was conducted, based on the CONSORT study protocol for randomized clinical trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0,2% CHX topical use (Experimental): Patients were asked to use topical medication containing 0,2% chlorhexidine 3 times a day, applying the size of a pea on the oral mucosa lesion until full wound healing or up to 14 days.
  Interventions: Drug: Chlorhexidine Gluconate
- 8,7% CHS topical use (Experimental): Patients were asked to use topical medication containing 8,7% choline salicylate 3 times a day, applying the size of a pea on the oral mucosa lesion until full wound healing or up to 14 days.
  Interventions: Drug: Choline Salicylate 8.7 % Oral Gel
- Control (Experimental): Patients were not using any topical medications.
  Interventions: Other: control group

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — topical preparation applied on oral mucosa lesion containing 0,2% CHX
  Arms: 0,2% CHX topical use
Drug: Choline Salicylate 8.7 % Oral Gel — topical preparation applied on oral mucosa lesion containing, ethanol-based
  Arms: 8,7% CHS topical use
Other: control group — no medication has been prescribed
  Arms: Control

SUMMARY:
The aim of the study was comparing the effectiveness of oral mucosa healing properties of different preparations: CHX=0,2% chorhexidine digluconate, CHS=8,7% choline salicylate, CON=control group, in patients with delivered removable dentures, during the adaptation period.

DETAILED DESCRIPTION:
The efficacy of oral topical medications in aiding regeneration and healing of oral soft mucosa, caused by the use of removable prosthetic restorations was analyzed. These medications, with different functional properties, are recommended for patients who develop oral mucosa lesions during adaptation to new removable prostheses. The evaluation of the efficacy of these agents was based on a comparison of the area of OML before and after the treatment. The study was designed to evaluate healing after the application of a topical medication containing 0.2% chlorhexidine digluconate and 8,7% choline salicylate as an active ingredient.

Patients were asked to use topical medication 3 times a day, applying the size of a pea on the oral mucosa lesion. Participants in groups CHX and CHS were instructed not to eat or drink for 1 hour following the application of medication because of its functional and antibacterial properties. Patients were asked to wear new dentures between control visits, even when they felt discomfort while using them. Patients in the control group were not using any topical medication. According to randomization patients suffering from oral mucosa lesion (OML) were divided into three groups.

Using a transparent millimeter grid superimposed on the OML, the Wound Surface Area (WSA) was measured in mm^2. A very precise measurement of the WSA was possible thanks to the use of a millimeter scale on the digital photo image. Every, even partially filled square was included in the area of the OML. Graphical analysis using Photo for Windows Software consisted of adding all the squares within which the OML was observed. All the intraoral images of OML have been taken in reproducible conditions (ambient light, lens and camera settings, distance 5 cm). This measurements were carried out during all check-up visits on day 0, 1, 4, 7 and 14.

ELIGIBILITY:
Inclusion Criteria:

* oral mucosa lesion OML as a result of new denture adaptation
* partial dentures II and III
* prostheses delivered for the during the period of the study patient
* patient consent

Exclusion Criteria:

* systemic conditions affecting the wound healing: diabetes
* prosthetic stomatitis according to Newton's classification
* parafunctional habits, bruxism
* autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Comparing the effectiveness of oral mucosa lesion healing of different preparations | From baseline assessment up to 2 weeks.
  Using a transparent millimeter grid superimposed on the oral mucosa lesion, the Wound Surface Area (WSA) was measured in mm^2.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of TMD Silesian Medical University, Zabrze, Poland